CLINICAL TRIAL: NCT00520325
Title: A Multi-Center Study of the Safety, Tolerability, Pharmacokinetics, and Dose Escalation of Intravenous Recombinant Human Mannose-Binding-Lectin (rhMBL) in MBL Deficient Pediatric Hematology/Oncology Patients With Fever and Neutropenia
Brief Title: A Study of Safety, Tolerability, and Pk of rhMBL in Pediatric Hematology/Oncology Pts With Fever and Neutropenia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor decision to terminate the study
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Responsible Party: Nazish Huq, Enzon Pharmaceuticals, Inc
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EZN-2232-03; NCI # 07-C-0027
Record Dates: First submitted 2007-08-23; First posted 2007-08-24 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2009-02

CONDITIONS: Cancer; Hematologic Diseases; Fever; Neutropenia
Keywords: MBL deficient oncologic hematologic pediatric fever neutropenia
MeSH Terms: conditions — Neoplasms; Hematologic Diseases; Fever; Neutropenia

ARMS (2):
- 0.5 mg/kg (Other)
  Interventions: Drug: Intravenous recombinant human mannose binding lectin
- 1.0 mg/kg (Other)
  Interventions: Drug: Intravenous recombinant human mannose binding lectin

INTERVENTIONS:
Drug: Intravenous recombinant human mannose binding lectin — Intravenous(i.v.) administration for one dose. Patients will be randomized to one of three cohorts: 0 mg/kg; 0.5 mg/kg, or 1.0 mg.kg
  Arms: 0.5 mg/kg
Drug: Intravenous recombinant human mannose binding lectin — Intravenous(i.v.) administration for one dose. Patients will be randomized to one of three cohorts: 0 mg/kg; 0.5 mg/kg, or 1.0 mg.kg
  Arms: 1.0 mg/kg

SUMMARY:
The goal of this clinical research study is to find the dose of EZN-2232 that can be given to MBL deficient pediatric cancer patients undergoing chemotherapy. The pharmacokinetics, pharmacodynamics, and safety of the study drug will also be studied.

DETAILED DESCRIPTION:
MBL deficient patients will be randomized in a ratio of 1:1 to receive a single dose of either 0.5 mg/kg or 1.0 mg/kg of intravenous rhMBL. A total of 24 patients will be treated in each of the rhMBL arms, (12 in the 0.5 mg/kg and 12 in the 1.0 mg/kg. All patients are to receive anti-infectious prophylactic supportive therapy as per institutional standards

ELIGIBILITY:
Inclusion Criteria: Patients must meet all of the following criteria to be eligible for enrollment into the study:

* Children ages 2 to 17 receiving chemotherapy for hematological/oncological diseases.
* Patients must have documented MBL levels <300 ng/mL in serum as evaluated in the screening protocol.
* Fever defined as an oral temperature equivalent of >100.4°F (38°C).
* Neutropenia defined as an absolute neutrophil count ≤1,000/mm3 with the anticipation that the counts will fall below 500/mm3.
* Receiving broad spectrum antibiotics for fever and neutropenia.
* Patients with age-adjusted normal serum creatinine OR a creatinine clearance >60 mL/min/1.73m2.
* Informed consent of the patient, parent or legally authorized representative obtained prior to entry.
* Reliable and willing to make themselves available for the duration of the study and to abide by the study restrictions.

Exclusion Criteria: Patients meeting any of the following exclusion criteria will not be eligible for enrollment.

* Patients receiving the preparative regimen for a bone marrow or hematopoietic stem cell transplantation.
* Concurrent serious illness in the opinion of the principal investigator that could potentially interfere with protocol compliance.
* Patient is pregnant, breast feeding or planning a pregnancy during the course of the study.
* Sexually active male and female patients not using an acceptable barrier method of contraception or practicing abstinence throughout the study and for at least 30 days after receiving their last treatment unless the patient is surgically or medically sterile.
* Patients with moderate or severe liver disease, as defined by:

AST or ALT >5 times upper limit of normal (ULN) OR Total bilirubin >2.5 times ULN.

* Patients with poor venous access that would preclude intravenous drug delivery or multiple blood draws.
* Current participation in another clinical study with an investigational agent and/or use of an investigational drug (not including investigational use of an FDA approved drug) in the 30 days before scheduled administration of rhMBL.
* Known allergic reactions to MBL or other human plasma products.
* Patients on hemodialysis unable to tolerate the volume of IV fluid on non-dialysis days.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Determine the safety and tolerability of intravenous rhMBL administered at dosages of 0.5 and 1.0 mg/kg to MBL deficient pediatric hematology/oncology patients during episodes of fever and neutropenia. | 1 month

SECONDARY OUTCOMES:
Determine the PK profile of intravenous rhMBL as a single dose escalation cohort design in MBL deficient pediatric oncology patients during episodes of fever and neutropenia. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Walsh, MD, Principal Investigator — NIH/National Cancer Institute